CLINICAL TRIAL: NCT00386347
Title: A Single Dose, Randomized, 5-Period, Balanced, Crossover Study to Assess the Relative Bioavailability of Three Formulations and Food Effect on GSK364735 and Pharmacokinetics Following a Double Blind, Placebo Controlled, Repeat Dose Administration to Healthy Subjects.
Brief Title: A Study To Evaluate Formulations And Food Effect On GSK364735 In Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GRZ108532
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infection; Infection, Human Immunodeficiency Virus
Keywords: HIV; repeat dose; pharmacokinetics; bioavailability; single-dose; food effect
MeSH Terms: conditions — HIV Infections; Infections; Acquired Immunodeficiency Syndrome | interventions — GSK364735

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK364735 oral solution and oral tablets

SUMMARY:
This study is a two-part study. Part one is designed to see how different formulations of GSK364735 are absorbed in the body and To see how food affects how GSK364735 is absorbed in the body. Part two is designed to see how repeat dosing affects how GSK364735 is absorbed in the body.

ELIGIBILITY:
Inclusion criteria:

* The subject is healthy with no clinically significant problems identified by the physician.
* Females of non-childbearing potential and males surgically sterile or agrees to birth control.
* Body mass Index (BMI) of 19-29.9 (kg/m2).

Exclusion criteria:

* As a result of the physical examination, lab results the Investigator considers the subject unfit for the study.
* Blood pressure and electrocardiogram is not normal
* A history of alcohol or illicit drug abuse.
* Tobacco use within 3 months.
* Positive for Hepatitis B surface antigen, Hepatitis C antibody or HIV antibody.
* Current use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements.
* Has participated in a clinical trial within 30 days prior to the first dose of study medication.
* Donated a pint of blood within a 56 day period.
* History of allergy to study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Start 2006-10

PRIMARY OUTCOMES:
Part 1: PK parameters Day 1: AUC(0-t), AUC(0-t), Cmax, and C12 and C24 Part 2: PK parameters on Day 6: AUC(0-t), Ct, and Cmax

SECONDARY OUTCOMES:
Part 1 and 2 safety measures: AE, Clinical labs, con meds, ECGs, and Vital signs Part 1: PK parameters Day 1: tmax, t1/2, tlag and CL/F Part 2: PK parameters Day 1&6: AUC 0-t, AUC 0-infinity, AUC 0-12, Cmax, C12 or C24, tmax, t1/2, CL/F, and tlag.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Evansville, Indiana, United States